CLINICAL TRIAL: NCT04803279
Title: Investigating Hearing With Ponto 3 SuperPower, a Bone Anchored Hearing Aid - Investigating Hear
Status: Completed | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC107
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss, Conductive; Hearing Loss Mixed; Hearing Disability; Conductive Hearing Loss; Ear Diseases; Conductive Hearing Loss, Bilateral; Conductive Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Ear Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ponto 3 SuperPower users: Patients who are fitted either unilaterally or bilaterally on abutment since the device came to the market in 2016, and who have followed the clinics normal routine fitting and follow up visits.
  They must also have undergone the normal procedures performed as part of the clinics routine for fitting and following up. Data was collected from these routine visits.
  Interventions: Device: Collection of Pure tone thresholds from audiogram measured prior to fitting of Ponto 3 SuperPower; Device: Collection of BC In-situ thresholds from BC In-situ audiogram measured during fitting of Ponto 3 SuperPower; Device: Collection of Aided sound field thresholds measured with the Ponto 3 SuperPower; Device: Collection of speech intelligibility scores; Device: Skin reaction; Device: Collection of Glasgow Benefit Inventory; Device: Collection of power-on usage time with Ponto 3 SuperPower

INTERVENTIONS:
Device: Collection of Pure tone thresholds from audiogram measured prior to fitting of Ponto 3 SuperPower — Unmasked and if available masked BC thresholds from audiogram obtained prior to Ponto 3 SuperPower were fitted.
Device: Collection of BC In-situ thresholds from BC In-situ audiogram measured during fitting of Ponto 3 SuperPower — BC In-situ thresholds will be collected from the BC In-situ audiogram obtained when Ponto 3 SuperPower were fitted
Device: Collection of Aided sound field thresholds measured with the Ponto 3 SuperPower — Sound field thresholds for frequencies 500Hz, 1kHz, 2 kHz, 3kHz and 4kHz will be collected from sound field audiogram obtained as follow-up after Ponto 3 SuperPower fitting, typically this is collected 3 months post fitting, alternatively from the fitting visit. Thresholds will be obtained aided, and when available unaided
Device: Collection of speech intelligibility scores — Speech intelligibility is measured in a sound treated room using sentence tests. The sentence tests used at Norwich and Norfolk hospital is the BKB (Bamford-Kowal-Bench) and/or the The AB[s] Isophonemic Monosyllabic Word test (7).
  The sentence tests are measured in quiet and/or with background speech-weighted noise.
Device: Skin reaction — Classification of skin reactions around skin penetrating implants will be made using the Holgers score. The Holgers classification is a scale from 0 to 4 that is used to grade skin reactions
Device: Collection of Glasgow Benefit Inventory — The Glasgow Benefit Inventory (GBI) contains 18 health status questions, which ask specific questions about how the health problem, in this study hearing loss, has affected their quality of life at the time the GBI is completed. In this study GBI has been collected on patients before intervention and 3 months after fitting of Ponto 3 SuperPower on abutment.
Device: Collection of power-on usage time with Ponto 3 SuperPower — Average power-on usage hours from Ponto 3 SuperPower will be collected.

SUMMARY:
The study is part of the Post Market Clinical Follow (PMCF) activity. The investigational device is the CE-marked Ponto 3 SuperPower (available on the market since December 2016) already fitted to the subjects, and data is collected retrospectively from clinical routine visits.

The study is a retrospective study. Therefore there will be no study visits for treatment or follow-up in the study.

Subject inclusion for this clinical investigation will be performed among subjects who has been fitted with the Ponto 3 SuperPower. To have a wide representative selection of subjects, enrollment will be spread over the 4 years since the device was available on the market since December 2016.

The endpoints in the study will investigate the improvement of hearing with the Ponto 3 SuperPower.

The data will be collected from the subjects in the time period from the clinical routine visit where the Ponto 3 SuperPower where fitted or just prior, and from the clinical routine visit following the fitting, where audiologic fitting follow-up procedures are performed (approximately 3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have consented to Section 3 of the document: "GDPR - what this means to you" (Appendix A) as part of a clinical routine visit.
2. Fitted unilaterally or bilaterally with the Ponto 3 SuperPower(s) on abutment(s)
3. Adult subjects (18 years or older)
4. Patient has attended a clinical routine visit where fitting of Ponto 3 SuperPower has been performed and at least one following clinical routine visit where audiological measurements has been performed

Exclusion Criteria:

There are no exclusion criteria in this study due to the retrospective nature of the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data collected from patients, who are Ponto 3 SuperPower users, and who have attended the Audiology Clinic at Norfolk and Norwich University Hospital (NNUH),Colney Ln, Norwich NR4 7UY, UK, in the period 2016-2020
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E FitzGerald, Bsc Phd, Principal Investigator — Norfolk & Norwich University Hospital NHS Foundation Trust
Locations (1):
- Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Target population 1 - Conductive/Mixed Hearing Loss (CHL/MHL) within indication Target population 1 - Bilaterally fitted CHL/MHL within indication Target population 2 - Single Sided Deafness (SSD) within indication
  Participants were assigned into groups based on type of hearing loss (not by ears or any other unit).
Groups:
- Target Population 1 - CHL/MHL: CHL/MHL within indication
- Target Population 2 - CHL/MHL Bilateral: Bilateral CHL/MHL within indication
- Target Population 3 - SSD: SSD within indication (TP3 - SSD)
Period: Overall Study
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - CHL/MHL Bilateral | Target Population 3 - SSD
Started | 46 | 8 | 3
Completed | 46 | 8 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Target Population 1 - CHL/MHL: TP 1 - Conductive Hearing Loss (CHL) / Mixed Hearing Loss (MHL) within indication.
- Target Population 2 - Bilateral: TP 2- Patients with CHL/MHL who were bilaterally fitted.
- Target Population 3 - SSD: TP 3 - Single Sided Deafness (SSD) within indication
- Total: Total of all reporting groups
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD | Total
Number analyzed (Participants) | 46 | 8 | 3 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (16.4) | 63.5 (15.6) | 57.7 (4.7) | 60.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 7 | 1 | 38
  Male | 16 | 1 | 2 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Gain Thresholds: Unaided Air Conduction (AC) Thresholds Compared to Aided Bone Conduction (BC) Thresholds, in Ponto 3 SuperPower Users With Conductive Hearing Loss (CHL) and/or Mixed Hearing Loss (MHL).
Description: Functional gain is the difference between the average unaided threshold measured across the frequencies of 500, 1000, 2000 and 4000 Hz and the average aided (i.e. with the Ponto 3 SuperPower) threshold measured across the frequencies of 500, 1000, 2000 and 4000 Hz.
  For bilaterally fitted patients, the best ear is selected.
Time Frame: Visit 2, 3 months
Population: Measurement not applicable for Target Population 3 - SSD
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Target Population 2 - Bilateral: TP 2 Patients with CHL/MHL who were bilaterally fitted.
- Target Population 3 - SSD: TP3 - Single Sided Deafness (SSD) within indication
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 46 | 8 | 0
dB
  Unaided AC [dB] | 70.2 (17.9) | 64.2 (19.4) |
  Aided sound field [dB]: number analyzed (Participants) | 33 | 7 | 0
  Aided sound field [dB] | 35.6 (9.0) | 35.2 (4.2) |
  Functional gain Unaided (AC) - Aided [dB]: number analyzed (Participants) | 33 | 7 | 0
  Functional gain Unaided (AC) - Aided [dB] | 36.0 (13.9) | 31.9 (15.4) |

2. Secondary Outcome: Functional Gain With the Ponto 3 SuperPower for Patients With CHL/MHL.
Description: Functional gain with Ponto 3 SuperPower, i.e. the difference between average unaided AC thresholds and aided sound field thresholds for frequencies 500, 1000, 2000, 3000 and 4000 Hz. For bilaterally fitted patients, the best ear is selected.
Time Frame: Visit 1, Day 1
Population: This variable is specific for patients with CHL/MHL only and thus not applicable for those with single-sided deafness, i.e., Target Population 3 - SSD.
Measure: Mean (Standard Deviation); unit: Functional gain Unaided (AC) - Aided [dB
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 46 | 8 | 0
Functional gain Unaided (AC) - Aided [dB
  500 Hz | 38.3 (17.6) | 35.0 (12.9) |
  1000 Hz | 37.4 (15.8) | 35.7 (15.7) |
  2000 Hz | 31.7 (17.1) | 26.4 (16.8) |
  3000 Hz | 34.2 (18.2) | 32.1 (24.5) |
  4000 Hz | 37.0 (16.5) | 35.0 (21.2) |

3. Secondary Outcome: Improvement of Speech Recognition in Quiet and in Noise With Ponto 3 SuperPower for Patients With CHL/MHL
Description: Aided speech recognition (% correct words) measured in quiet and in noise with the BKB sentence test and the AB[s] short list test averaged across patients. Only participants with data for both visits were included in analysis.
Time Frame: Visit 2, 3 months
Population: Participants with speech recognition scores recorded included in analysis speech recognition scores. This variable is specific for patients with CHL/MHL only and thus not applicable for those with single-sided deafness, i.e., Target Population 3 - SSD.
Measure: Mean (Standard Deviation); unit: percent correct words
Groups:
- Target Population 3 - SSD: TP3 - Single Sided Deafness (SSD) within population
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 46 | 8 | 0
percent correct words
  BKB Sentence Test in Noise: number analyzed (Participants) | 14 | 7 | 0
  BKB Sentence Test in Noise | 73.5 (19.0) | 66.5 (23.8) |
  BKB Sentence Test in Quiet: number analyzed (Participants) | 18 | 7 | 0
  BKB Sentence Test in Quiet | 88.6 (11.3) | 91.5 (7.1) |
  AB[s] short list in Noise: number analyzed (Participants) | 33 | 7 | 0
  AB[s] short list in Noise | 67.6 (21.0) | 59.0 (21.8) |
  AB[s] short list in Quiet: number analyzed (Participants) | 38 | 7 | 0
  AB[s] short list in Quiet | 84.1 (18.7) | 87.7 (9.3) |

4. Secondary Outcome: Speech Recognition in Noise Improvements With Ponto 3 SuperPower on for Patients With SSD
Description: Difference in speech recognition score (%) for speech recognition in noise between unaided and aided when speech is directed to the aided ear, and noise is directed to the non-implanted ear, and when speech is directed to the non-implanted ear, and when noise is directed to the aided ear.
  Aided and unaided speech recognition (% correct words) measured with the AB[s] short list.
Time Frame: Visit 2, 3 months
Population: The aided condition was obtained from two patients while the unaided condition was measured for one patient from the SSD patients within indication (TP2 - SSD, n=3). This outcome is only applicable for Target Population 3 - SSD.
Measure: Mean (Standard Deviation); unit: percent correct words
Groups:
- Target Population 1 - CHL/MHL: TP1 - Conductive Hearing Loss (CHL)/Mixed Hearing Loss (MHL) within indication
- Target Population 2 - Bilateral: TP2 - Patients with CHL/MHL who were bilaterally fitted
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 0 | 0 | 3
percent correct words
  Aided SimplatedNnon-implanted - % correct: number analyzed (Participants) | 0 | 0 | 2
  Aided SimplatedNnon-implanted - % correct |  |  | 60.0 (9.5)
  Unaided SimplatedNnon-implanted - % correct: number analyzed (Participants) | 0 | 0 | 1
  Unaided SimplatedNnon-implanted - % correct |  |  | 36.7 (0)
  Difference: Aided - Unaided SimplatedNnon-implanted - % correct: number analyzed (Participants) | 0 | 0 | 1
  Difference: Aided - Unaided SimplatedNnon-implanted - % correct |  |  | 30.0 (0)
  Aided Snon-implatedNimplanted - % correct: number analyzed (Participants) | 0 | 0 | 2
  Aided Snon-implatedNimplanted - % correct |  |  | 80.0 (23.6)
  Unaided Snon-implatedNimplanted - % correct: number analyzed (Participants) | 0 | 0 | 1
  Unaided Snon-implatedNimplanted - % correct |  |  | 91.3 (0)
  Difference: Aided- Unaided Snon-implatedNimplanted - % correct: number analyzed (Participants) | 0 | 0 | 1
  Difference: Aided- Unaided Snon-implatedNimplanted - % correct |  |  | 5.40 (0)

5. Secondary Outcome: Degree of Compensation for Hearing Loss on the Implanted Ear(s) With the Ponto 3 SuperPower for Patients With CHL/MHL.
Description: Effective gain with Ponto 3 SuperPower, i.e. the difference between aided sound field thresholds and the BC In-situ thresholds on the aided ear(s) measured when the Ponto 3 SuperPower(s) was fitted. The effective gain is calculated as the average (PTA4) of frequencies 500, 1000, 2000 and 4000 Hz. Only participants with data for both study visits were included in the analysis.
Time Frame: visit 2, 3 months
Population: Analysis includes tested frequencies. This variable is specific for patients with CHL/MHL only and thus not applicable for those with single-sided deafness, i.e., Target Population 3 - SSD.
Measure: Mean (Standard Deviation); unit: Effective gain Aided - BC In-situ [dB]
Groups:
- Target Population 2 - SSD: TP3 - Single Sided Deafness (SSD) within indication
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 2 - SSD
Number analyzed (Participants) | 46 | 8 | 0
Effective gain Aided - BC In-situ [dB]
  PTA 4: number analyzed (Participants) | 33 | 7 | 0
  PTA 4 | -0.22 (7.96) | -0.36 (8.5) |
  500 Hz: number analyzed (Participants) | 33 | 7 | 0
  500 Hz | 4.09 (9.88) | 5.71 (8.38) |
  1000 Hz: number analyzed (Participants) | 33 | 7 | 0
  1000 Hz | -2.42 (10.01) | -2.14 (8.59) |
  2000 Hz: number analyzed (Participants) | 33 | 7 | 0
  2000 Hz | -0.46 (9.95) | -1.43 (11.07) |
  3000 Hz: number analyzed (Participants) | 31 | 7 | 0
  3000 Hz | 1.45 (9.68) | -0.71 (9.76) |
  4000 Hz: number analyzed (Participants) | 32 | 7 | 0
  4000 Hz | -2.03 (9.74) | -3.57 (12.82) |

6. Secondary Outcome: Quality of Life Improvements With the Ponto 3 SuperPower
Description: Glasgow Benefit Inventory (GBI) total score per target population.
  The GBI consists of 18 items, each on a 5 point Likert scale. Responses are scaled and averaged to give a score with a range -100 (poorest outcome) through 0 (no change) to +100 (best outcome).
Time Frame: Visit 2, 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Target Population 1- CHL/MHL: CHL/MHL within indication. Only participants with recorded GBI scores are analyzed.
- Target Population 2 - Bilateral: Bilateral CHL/MHL within indication
Arm/Group | Target Population 1- CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 46 | 8 | 3
units on a scale | 53.9 (20.9) | 56.4 (26.6) | 41.9 (24.3)

7. Secondary Outcome: Individual Level Evaluation of Objectives 1-6; Improved Hearing
Description: Improved hearing was analyzed as the percentage of subjects whose performance is better or equal in the unaided to aided comparisons, i.e., have a difference ≥0.
  Functional gain was used for CHL/MHL patients and speech recognition in noise was used for SSD patients.
Time Frame: Change between visit 1 (day 1) and visit 2 (3 months)t of study
Population: Functional gain for CHL/MHL based on PTA4 was not available for all individuals. Speech recognition in noise was measured aided and unaided for only one SSD patient within indication (TP3 - SSD).
Measure: Count of Participants; unit: Participants
Groups:
- Target Group 2 - Bilateral: Bilateral CHL/MHL within indication
Arm/Group | Target Population 1 - CHL/MHL | Target Group 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 33 | 7 | 1
Participants | 33 | 7 | 1

8. Secondary Outcome: Air to Bone Gap (PTA3) on the Implanted Ear(s) for Patients With CHL/MHL
Description: The difference between masked (if not available unmasked) BC and AC thresholds (unaided), denoted 'air to bone gap', calculated for frequencies 500, 1000, and 2000 Hz for the patients with CHL/MHL within indication on the implanted ear. For bilateral patients, the best ear was selected. Only participants that had complete data for these frequencies were included in the analysis.
Time Frame: Visit 1 day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Air to bone gap AC - BC [dB]
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 46 | 8 | 0
Air to bone gap AC - BC [dB]
  PTA3: number analyzed (Participants) | 38 | 3 | 0
  PTA3 | 33.6 (12.4) | 21.7 (16.7) |
  500 Hz: number analyzed (Participants) | 37 | 3 | 0
  500 Hz | 37.7 (17.9) | 25.0 (18.0) |
  1000 Hz: number analyzed (Participants) | 38 | 3 | 0
  1000 Hz | 37.4 (13.1) | 30.0 (20.0) |
  2000 Hz: number analyzed (Participants) | 35 | 3 | 0
  2000 Hz | 25.7 (13.1) | 15.0 (14.1) |

9. Secondary Outcome: Skin Condition Assessment Around the Abutment
Description: Skin condition around the abutment was assessed via Holgers score (scale 0-4).
  Holgers 0: No skin reaction Holgers 1: Redness with slight swelling Holgers 2: Redness, moistness, and moderate swelling Holgers 3: Redness, moistness, and moderate swelling with tissue granulation Holgers 4: Profound signs of infection, resulting in removal of the implant
  Only participants who had recorded Holgers score in record were analyzed.
Time Frame: Visit 2, 3 months
Population: For Target Population 2 - Bilateral both treated ears are considered.
Measure: Count of Units; unit: Number of ears
Units Other Than Participants: Number of ears
Arm/Group | Target Population 1 - CHL/MHL | Target Population 2 - Bilateral | Target Population 3 - SSD
Number analyzed (Participants) | 36 | 8 | 2
Number analyzed (Number of ears) | 36 | 16 | 2
Number of ears
  Holger's score 0-1 | 35 | 15 | 2
  Holger's score 2-4 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Not applicable due to the retrospective nature of the study.
Description: Not applicable due to the retrospective nature of the study.
Groups:
- All Enrolled Participants: Existing Ponto 3 SuperPower users who were fitted either unilaterally or bilaterally on abutment since the device came to the market in 2016, and who have followed the clinics normal routine fitting and follow up visits.
  The adverse events are reported for all participants as a single group rather than by the analysis groups, primarily as this was a retrospective study design and furthermore one would not expect differences in hearing loss etiology (again, the analysis groups) would result in differences in adverse events in this retrospective study.
Arm/Group | All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/79/NCT04803279/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT04803279/SAP_001.pdf